CLINICAL TRIAL: NCT06960889
Title: A Retrospective Clinical Study Exploring Prognostic Factors in Esophageal Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-163
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Esophageal Cancer (EsC)
Keywords: Prognostic factors; Treatment strategies; Efficacy comparison; Esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy; Immunotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Radiotherapy Group: Participants will receive definitive radiotherapy or radiotherapy-based combined modality therapy.
  Interventions: Other: radiotherapy
- Immunotherapy Group: Participants will receive immune checkpoint inhibitors as monotherapy or in combination with other therapies.
  Interventions: Drug: Immunotherapy
- Surgery Group: Participants will undergo radical esophagectomy with or without neoadjuvant/adjuvant therapy.
  Interventions: Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines

INTERVENTIONS:
Other: radiotherapy — Definitive radiotherapy or radiotherapy-based combined modality therapy
  Groups: Radiotherapy Group
Drug: Immunotherapy — Immune checkpoint inhibitors as monotherapy or in combination with other therapies
  Groups: Immunotherapy Group
Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines — Radical esophagectomy with or without neoadjuvant/adjuvant therapy
  Groups: Surgery Group

SUMMARY:
This single-center, retrospective, 7-year observational study aims to investigate prognostic factors in esophageal cancer patients. Adults (≥18 years) with histologically confirmed esophageal cancer who received antitumor therapy between January 2017 and December 2024 were consecutively enrolled. Patient-level data (clinical characteristics, routine laboratory tests, tumor information, and treatment details) were retrospectively collected from electronic medical records to analyze key factors influencing treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Waiver of informed consent for deceased or lost-to-follow-up patients (January 2017-March 2024)
2. Voluntary signed informed consent from surviving patients who could be contacted
3. Treatment at Nanfang Hospital, Southern Medical University (January 2017-December 2024)
4. Received antitumor therapy for esophageal cancer
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2

Exclusion Criteria:

1. Concurrent other malignancies
2. Patients deemed ineligible by investigators

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Esophageal Cancer Patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From the date of treatment initiation to the date of death from any cause,assessed up to 120 months.
  The length of time from the start of treatment until death from any cause, evaluating the long-term survival benefit of the combined therapy.

SECONDARY OUTCOMES:
Pathologic Complete Response ( pCR ) | Perioperative
  The absence of residual viable tumor cells in both the primary esophageal tumor and regional lymph nodes after completion of surgery, indicating a complete pathological response.
Major Pathological Response Rate (MPR) | Perioperative
  The proportion of patients with ≤10% residual viable tumor cells in resected specimens
Progression-Free Survival (PFS) | From treatment initiation to disease progression or death, assessed up to 100 months
  The duration from treatment start until radiologically confirmed disease progression (per RECIST v1.1) or death from any cause, evaluating therapeutic efficacy in delaying tumor growth.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shi X, Zhao H, Yu J, Cai P, Zhou S, Yang N, Li D. Changes in PD-1 expression on T lymphocyte subsets and related immune indicators before and after definitive chemoradiotherapy for esophageal squamous cell carcinoma. Ann Med. 2025 Dec;57(1):2445190. doi: 10.1080/07853890.2024.2445190. Epub 2024 Dec 23. PMID 39713872
- [Background] Lin FC, Chang WL, Chiang NJ, Lin MY, Chung TJ, Pao TH, Lai WW, Tseng YL, Yen YT, Sheu BS. Radiation dose escalation can improve local disease control and survival among esophageal cancer patients with large primary tumor volume receiving definitive chemoradiotherapy. PLoS One. 2020 Aug 6;15(8):e0237114. doi: 10.1371/journal.pone.0237114. eCollection 2020. PMID 32760099
- [Background] Dong J, Li C, Wang B, Li Y, Wang S, Cui H, Gao M. Prognostic analysis of esophageal cancer patients after neoadjuvant therapy. Front Immunol. 2025 Feb 21;16:1553086. doi: 10.3389/fimmu.2025.1553086. eCollection 2025. PMID 40061941
- [Background] Yang H, Liu H, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Chen Z, Yang H, Wang J, Pang Q, Zheng X, Yang H, Li T, Lordick F, D'Journo XB, Cerfolio RJ, Korst RJ, Novoa NM, Swanson SJ, Brunelli A, Ismail M, Fernando HC, Zhang X, Li Q, Wang G, Chen B, Mao T, Kong M, Guo X, Lin T, Liu M, Fu J; AME Thoracic Surgery Collaborative Group. Neoadjuvant Chemoradiotherapy Followed by Surgery Versus Surgery Alone for Locally Advanced Squamous Cell Carcinoma of the Esophagus (NEOCRTEC5010): A Phase III Multicenter, Randomized, Open-Label Clinical Trial. J Clin Oncol. 2018 Sep 20;36(27):2796-2803. doi: 10.1200/JCO.2018.79.1483. Epub 2018 Aug 8. PMID 30089078
- [Background] Wang ZX, Cui C, Yao J, Zhang Y, Li M, Feng J, Yang S, Fan Y, Shi J, Zhang X, Shen L, Shu Y, Wang C, Dai T, Mao T, Chen L, Guo Z, Liu B, Pan H, Cang S, Jiang Y, Wang J, Ye M, Chen Z, Jiang D, Lin Q, Ren W, Wang J, Wu L, Xu Y, Miao Z, Sun M, Xie C, Liu Y, Wang Q, Zhao L, Li Q, Huang C, Jiang K, Yang K, Li D, Liu Y, Zhu Z, Chen R, Jia L, Li W, Liao W, Liu HX, Ma D, Ma J, Qin Y, Shi Z, Wei Q, Xiao K, Zhang Y, Zhang Y, Chen X, Dai G, He J, Li J, Li G, Liu Y, Liu Z, Yuan X, Zhang J, Fu Z, He Y, Ju F, Liu Z, Tang P, Wang T, Wang W, Zhang J, Luo X, Tang X, May R, Feng H, Yao S, Keegan P, Xu RH, Wang F. Toripalimab plus chemotherapy in treatment-naive, advanced esophageal squamous cell carcinoma (JUPITER-06): A multi-center phase 3 trial. Cancer Cell. 2022 Mar 14;40(3):277-288.e3. doi: 10.1016/j.ccell.2022.02.007. Epub 2022 Mar 3. PMID 35245446
- [Background] Lu Z, Wang J, Shu Y, Liu L, Kong L, Yang L, Wang B, Sun G, Ji Y, Cao G, Liu H, Cui T, Li N, Qiu W, Li G, Hou X, Luo H, Xue L, Zhang Y, Yue W, Liu Z, Wang X, Gao S, Pan Y, Galais MP, Zaanan A, Ma Z, Li H, Wang Y, Shen L; ORIENT-15 study group. Sintilimab versus placebo in combination with chemotherapy as first line treatment for locally advanced or metastatic oesophageal squamous cell carcinoma (ORIENT-15): multicentre, randomised, double blind, phase 3 trial. BMJ. 2022 Apr 19;377:e068714. doi: 10.1136/bmj-2021-068714. PMID 35440464
- [Background] Li QQ, Liu MZ, Hu YH, Liu H, He ZY, Lin HX. Definitive concomitant chemoradiotherapy with docetaxel and cisplatin in squamous esophageal carcinoma. Dis Esophagus. 2010 Apr;23(3):253-9. doi: 10.1111/j.1442-2050.2009.01003.x. Epub 2009 Aug 28. PMID 19732130
- [Background] Chen Y, Ye J, Zhu Z, Zhao W, Zhou J, Wu C, Tang H, Fan M, Li L, Lin Q, Xia Y, Li Y, Li J, Jia H, Lu S, Zhang Z, Zhao K. Comparing Paclitaxel Plus Fluorouracil Versus Cisplatin Plus Fluorouracil in Chemoradiotherapy for Locally Advanced Esophageal Squamous Cell Cancer: A Randomized, Multicenter, Phase III Clinical Trial. J Clin Oncol. 2019 Jul 10;37(20):1695-1703. doi: 10.1200/JCO.18.02122. Epub 2019 Mar 28. PMID 30920880
- [Background] Lockhart AC, Reed CE, Decker PA, Meyers BF, Ferguson MK, Oeltjen AR, Putnam JB, Cassiv SD, Montero AJ, Schefter TE. Phase II study of neoadjuvant therapy with docetaxel, cisplatin, panitumumab, and radiation therapy followed by surgery in patients with locally advanced adenocarcinoma of the distal esophagus (ACOSOG Z4051). Ann Oncol. 2019 Feb 1;30(2):345. doi: 10.1093/annonc/mdx813. No abstract available. PMID 29390067
- [Background] Eyck BM, van Lanschot JJB, Hulshof MCCM, van der Wilk BJ, Shapiro J, van Hagen P, van Berge Henegouwen MI, Wijnhoven BPL, van Laarhoven HWM, Nieuwenhuijzen GAP, Hospers GAP, Bonenkamp JJ, Cuesta MA, Blaisse RJB, Busch OR, Creemers GM, Punt CJA, Plukker JTM, Verheul HMW, Spillenaar Bilgen EJ, van der Sangen MJC, Rozema T, Ten Kate FJW, Beukema JC, Piet AHM, van Rij CM, Reinders JG, Tilanus HW, Steyerberg EW, van der Gaast A; CROSS Study Group. Ten-Year Outcome of Neoadjuvant Chemoradiotherapy Plus Surgery for Esophageal Cancer: The Randomized Controlled CROSS Trial. J Clin Oncol. 2021 Jun 20;39(18):1995-2004. doi: 10.1200/JCO.20.03614. Epub 2021 Apr 23. PMID 33891478
- [Background] Yang H, Liu H, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Chen Z, Yang H, Wang J, Pang Q, Zheng X, Yang H, Li T, Zhang X, Li Q, Wang G, Chen B, Mao T, Kong M, Guo X, Lin T, Liu M, Fu J. Long-term Efficacy of Neoadjuvant Chemoradiotherapy Plus Surgery for the Treatment of Locally Advanced Esophageal Squamous Cell Carcinoma: The NEOCRTEC5010 Randomized Clinical Trial. JAMA Surg. 2021 Aug 1;156(8):721-729. doi: 10.1001/jamasurg.2021.2373. PMID 34160577
- [Background] Biere SS, van Berge Henegouwen MI, Maas KW, Bonavina L, Rosman C, Garcia JR, Gisbertz SS, Klinkenbijl JH, Hollmann MW, de Lange ES, Bonjer HJ, van der Peet DL, Cuesta MA. Minimally invasive versus open oesophagectomy for patients with oesophageal cancer: a multicentre, open-label, randomised controlled trial. Lancet. 2012 May 19;379(9829):1887-92. doi: 10.1016/S0140-6736(12)60516-9. Epub 2012 May 1. PMID 22552194
- [Background] Kwon Y, Yun JK, Jeon YH, Kim YH. Long-term oncologic outcomes of robot-assisted versus conventional open esophagectomy for esophageal cancer: Propensity-score matched anaylsis. Eur J Surg Oncol. 2025 May;51(5):109591. doi: 10.1016/j.ejso.2025.109591. Epub 2025 Jan 9. PMID 39808888
- [Background] Filho AM, Laversanne M, Ferlay J, Colombet M, Pineros M, Znaor A, Parkin DM, Soerjomataram I, Bray F. The GLOBOCAN 2022 cancer estimates: Data sources, methods, and a snapshot of the cancer burden worldwide. Int J Cancer. 2025 Apr 1;156(7):1336-1346. doi: 10.1002/ijc.35278. Epub 2024 Dec 17. PMID 39688499